CLINICAL TRIAL: NCT01573962
Title: A Sample Collection Study to Validate the Astute Medical NephroCheck Test in Critically Ill Subjects at Risk for Acute Kidney Injury
Status: Completed | Type: Observational
Sponsor: Astute Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Topaz
Record Dates: First submitted 2012-04-06; First posted 2012-04-10 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2013-09

CONDITIONS: Acute Kidney Injury
Keywords: Kidney Renal
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this sample collection study is to collect blood and urine samples. This study is observational and will have no impact on the medical management of the subject.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 21 years of age or older
* Subjects must be enrolled (first study-specific sample collection) within 24 hours of ICU admission
* Subjects enrolled from ED or Floor must be admitted to the ICU within 24 hours of enrollment
* Subjects enrolled in the ICU must have been admitted to the ICU or transferred into the study ICU from another ICU no more than 24 hours prior to enrollment
* Expected to remain in the ICU for at least 48 hours after enrollment
* Use of indwelling urinary catheter as standard care expected for at least 48 hours after enrollment
* At least one of the following acute conditions documented within 24 hours prior to enrollment
* Respiratory SOFA score of ≥ 2 (PaO2/FiO2 <300)
* Cardiovascular SOFA score of ≥ 1 (MAP < 70 mm Hg and/or any vasopressor required
* Subject (or authorized representative) able and willing to provide written informed consent for study participation.

Exclusion Criteria:

* Special populations including women with known pregnancy, prisoners or institutionalized individuals
* Previous renal transplantation
* Known moderate to severe AKI prior to enrollment (e.g., RIFLE-I or RIFLE-F/ AKIN 2 or AKIN 3
* Already receiving dialysis (either acute or chronic) or in imminent need of dialysis at the time of enrollment
* Known infection with human immunodeficiency virus (HIV) or active hepatitis (acute or chronic)
* Subjects with a history of Chronic Kidney Disease (CKD) without a baseline serum creatinine value (baseline within 6 months of enrollment)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients at risk of AKI.
Sampling Method: Non-Probability Sample
Enrollment: 420 (Actual)
Dates: Start 2012-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
A Sample Collection Study to Validate the Astute Medical NephroCheck Test in Critically Ill Subjects at Risk for Acute Kidney Injury | 04/1/2012 to 3/29/13

CONTACTS AND LOCATIONS:
Overall Officials: John Kellum, Ph.D., Principal Investigator — Professor, Critical Care Medicine, University of Pittsburgh
Locations (21):
- United States (21):
  - Loma Linda, California
  - Los Angels, California
  - Washington D.C., District of Columbia
  - Gainesville, Florida
  - Tampa, Florida
  - Idaho Falls, Idaho
  - Chicago, Illinois
  - Shreveport, Louisiana
  - Baltimore, Maryland
  - Ann Arbor, Michigan
  - Minneapolis, Minnesota
  - Missoula, Montana
  - Rochester, New York
  - The Bronx, New York
  - Durham, North Carolina
  - Akron, Ohio
  - Portland, Oregon
  - Pittsburgh, Pennsylvania
  - Nashville, Tennessee
  - Houston, Texas
  - Richmond, Virginia

REFERENCES:
- [Derived] Bihorac A, Chawla LS, Shaw AD, Al-Khafaji A, Davison DL, Demuth GE, Fitzgerald R, Gong MN, Graham DD, Gunnerson K, Heung M, Jortani S, Kleerup E, Koyner JL, Krell K, Letourneau J, Lissauer M, Miner J, Nguyen HB, Ortega LM, Self WH, Sellman R, Shi J, Straseski J, Szalados JE, Wilber ST, Walker MG, Wilson J, Wunderink R, Zimmerman J, Kellum JA. Validation of cell-cycle arrest biomarkers for acute kidney injury using clinical adjudication. Am J Respir Crit Care Med. 2014 Apr 15;189(8):932-9. doi: 10.1164/rccm.201401-0077OC. PMID 24559465